CLINICAL TRIAL: NCT03705507
Title: International Phase I/II Expansion Trial of the MEK Inhibitor Selumetinib in Combination With Dexamethasone for the Treatment of Relapsed/Refractory RAS-pathway Mutated Paediatric and Adult Acute Lymphoblastic Leukaemia
Brief Title: International Trial of Selumetinib in Combination With Dexamethasone for the Treatment of Acute Lymphoblastic Leukaemia
Acronym: SeluDex
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor recruitment, due to a change in the standard of care for this patient population with the use of CAR-T cells
Sponsor: University of Birmingham (Other)
Collaborators: Cancer Research UK (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_16-186; 2016-003904-29 (EudraCT Number); ISRCTN92323261 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2018-07-04; First posted 2018-10-15 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia, Adult; Acute Lymphoblastic Leukemia, Pediatric; Acute Lymphoblastic Leukemia, in Relapse; Acute Lymphoblastic Leukemia Recurrent
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — AZD 6244; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Group P will enrol all patients under 18 years of age and Group A will enrol all patients who are 18 years or older.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selumetinib + Dexamethasone - Group A (18 years and above) (Experimental): Patients will receive the adult cohort specified dose of selumetinib by mouth, as a single dose on cycle 1 day 1, then twice daily continuously from cycle 1 day 4 onwards. Combined with pulsed doses of dexamethasone at 6mg/m2/day on days 2-4 and 8-11 then at 4mg/m2/day on days 15-18 and 22-25 divided into two doses (as per local practice) by mouth during cycle 1, then on days 1-4 at 4mg/m2/day at the start of cycle 2, then on days 1-5 at 6mg/m2/day during subsequent cycles.
  Interventions: Drug: Selumetinib; Drug: Dexamethasone
- Selumetinib + Dexamethasone - Group P (under 18 years) (Experimental): Patients will receive the paediatric cohort specified dose of selumetinib by mouth, as a single dose on cycle 1 day 1, then twice daily continuously from cycle 1 day 4 onwards. Combined with pulsed doses of dexamethasone at 6mg/m2/day on days 2-4 and 8-11 then at 4mg/m2/day on days 15-18 and 22-25 divided into two doses (as per local practice) by mouth during cycle 1, then on days 1-4 at 4mg/m2/day at the start of cycle 2, then on days 1-5 at 6mg/m2/day during subsequent cycles.
  Interventions: Drug: Selumetinib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selumetinib — Selumetinib is a small molecule inhibitor of the MEK protein
  Other Names: AZD6244
Drug: Dexamethasone — Steroid used for the treatment and management of a number of conditions including cancers and leukaemias.

SUMMARY:
This trial is to investigate the combination of selumetinib and dexamethasone in the treatment of acute lymphoblastic leukaemia (ALL) in both adults and children. Phase I is to find the most suitable dose of selumetinib to safely give with dexamethasone. Phase II will use this dose to find out how well the combination works.

DETAILED DESCRIPTION:
Acute lymphoblastic leukaemia (ALL) is the most common childhood cancer worldwide. The overall newly diagnosed ALL cure rate is approaching 90% however children with relapsed ALL often do not survive. The frequency of ALL in adults is significantly lower however more challenging to treat compared to childhood ALL. Adult ALL is more resistant to chemotherapy and patient have reduced treatment tolerance (particularly the elderly population) therefore overall survival rates are low. Therefore there is a need to develop more effective treatment which improves survival rates for this patient population.

Those eligible in the paediatric setting are in their second or further relapse, often after a previous allogeneic stem cell transplant (SCT), and usually in a palliative situation. Adult patients who are not suitable for more intensive therapy can enter the trial in first relapse. The trial offers an out-patient based treatment approach of this heavily pre-treated patient group. The trial includes patients with B-cell precursor and T-ALL irrespective of Central Nervous System (CNS) disease status.CNS positive patients and patients with T-ALL are usually excluded from other early phase clinical trials. If treatment is successful, patients could continue with other therapies/trials once complete remission achieved (e.g. Chimeric Antigen Receptor (CAR) T cell therapy).

Selumetinib is a small molecule inhibitor of MEK, a protein in the RAS-pathway. Mutations in genes in the RAS pathway have been found in a large proportion of patients with ALL. Selumetinib targets this over-activated pathway to arrest cancer cell growth. Dexamethasone is a steroid important in the treatment of leukaemia to stimulate the death of cancer cells. The SeluDex trial is for patients with relapsed or refractory RAS-pathway mutated ALL.

The primary objective of this trial in Phase I is to see what dose of selumetinib can safely be given in combination with dexamethasone in participants. During Phase II, the primary objective is to assess the preliminary information regarding the effectiveness of this combined treatment.

ELIGIBILITY:
Inclusion Criteria:

* Morphologically proven relapsed/refractory (M2 or M3 marrow; ≥1st relapse for adults, ≥2nd relapse in paediatric group - see Protocol Appendix 5) or progressive B cell precursor or T-Acute Lymphoblastic Leukaemia (ALL) with demonstrated RAS pathway activating mutations (NRAS, KRAS, FLT3, PTPN11, cCBL, NF1, BRAF, IKZF2, IKZF3, IL7Rα or JAK1) identified during the trial screening process
* B cell precursor patients must either:

  * Have received CAR -T cell therapy, or
  * Be awaiting CAR -T cell therapy, or
  * Be considered ineligible for CAR -T cell therapy
* Group P (paediatric): <18 years of age; Group A (adult): ≥18 years of age
* Adequate renal function:

  * Group A: Serum creatinine <1.5 x upper limit of normal (ULN)
  * Group P as follows:

    * 5 years: Serum creatinine <0.8 mg/dL or 70 μmol/L, > 5 years but ≤ 10 years: Serum creatinine <1 mg/dL or 88 μmol/L, > 10 years but ≤ 15 years: Serum creatinine <1.2 mg/dL or 106 μmol/L, > 15 years: Serum creatinine <1.5 mg/dL or 132 μmol/L
* Patient is able to swallow selumetinib capsules whole
* Performance status (PS): Group A - Eastern Cooperative Oncology Group (ECOG) ≤2 (Protocol Appendix 6); Group P - Lansky play scale ≥60% (Protocol Appendix 7) or Karnofsky scale ≥60% (Appendix 8)
* Women of childbearing potential (see protocol section 7.9.3 for definition) must have a negative pregnancy test
* Patients who are women of childbearing potential and male patients with partners who are women of childbearing potential must agree to use appropriate contraception (see protocol section 7.9.3 for definition) whilst on trial
* Written informed consent
* Absence of any psychological, familial, sociological or geographical factors potentially hampering compliance with the trial protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Patients who relapse or progress after Haematopoetic Stem Cell Transplant (HSCT) need to be at least at day +100, with no signs of Graft versus Host Disease and off immunosuppressive therapy for at least one week.
* Patients who relapse or progress after CAR T cell therapy should be at least 4 weeks after infusion of CAR T cells.
* Patients must have a body surface area (BSA) ≥ 0.55 m2.

Exclusion Criteria:

* ALL without presence of RAS-pathway activating mutations
* Mature B-cell leukaemia and Philadelphia positive ALL
* Prior exposure to MEK, RAS or RAF inhibitors
* Any unresolved toxicity ≥ CTCAE Grade 2 from previous anti-cancer therapy, except for alopecia
* Cardiac conditions as follows:

Group A and P

* Prior or current cardiomyopathy including but not limited to the following:

  * Known hypertrophic cardiomyopathy
  * Known arrhythmogenic right ventricular cardiomyopathy
* Even if full recovery has occurred, previous moderate or severe impairment of left ventricular systolic function (LVEF <45% on Echocardiogram (ECHO) in Group A; SF <29% in Group P but excluding transient impairments due to e.g. anaemia/sepsis or results not thought to represent a true reflection of cardiac function)
* Severe valvular heart disease
* Severe congenital heart disease
* Uncontrolled hypertension:

  * Group A: BP ≥150/95 mmHg despite medical therapy
  * Group P: BP ≥95th percentile for age, height and gender (please refer to Blood Pressure by Age and Height Percentiles tables in Protocol Appendices 8 and 9) Group A
* Baseline (LVEF) below the lower limit of normal (LLN) or <55% measured by ECHO
* Acute coronary syndrome within 6 months prior to trial registration
* Uncontrolled Angina - Canadian Cardiovascular Society grade II-IV despite medical therapy (Protocol Appendix 11)
* Symptomatic heart failure New York Heart Association (NYHA) Class II-IV, prior or current cardiomyopathy, or severe valvular heart disease (Protocol Appendix 12)
* Atrial fibrillation with a ventricular rate >100 bpm on Electrocardiogram (ECG) at rest
* QTcF >450ms in male patients or ≥460ms in female patients, or other factors that increase the risk of QT prolongation Group P
* Baseline SF <29%
* Atrial fibrillation with a ventricular rate >130 bpm on Electrocardiogram (ECG) at rest
* QTcF >450ms in patients <12 years or ≥460ms in patients ≥12 but <18 years
* Ophthalmological conditions as follows:

  * Current or past history of retinal pigment epithelial detachment (RPED)/central serous retinopathy (CSR) or retinal vein occlusion (RVO)
  * Intraocular pressure (IOP) > 21 mmHg or uncontrolled glaucoma (irrespective of IOP)
* Pregnant and breast feeding females
* Known severe hypersensitivity to selumetinib, dexamethasone or combination medications or any excipient of these medicinal products, or history of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib
* Have received or are receiving an Investigational Medicinal Product (IMP) or other systemic anti-cancer treatment (not including dexamethasone, prednisolone or hydroxycarbamide) within 4 weeks (6 weeks for nitrosoureas, mitomycin, and suramin) prior to trial registration, or within a period during which the IMP or systemic anticancer treatment has not been cleared from the body (e.g. a period of 5 'half-lives'), whichever is the most appropriate and as judged by the investigator
* Have had recent major surgery within a minimum 4 weeks prior to trial registration, with the exception of surgical placement of vascular access
* Have received radiation therapy within 4 weeks prior to trial registration, or limited field of radiation for palliation within 7 days of the first dose of trial treatment
* Laboratory values as listed below (SI units):

  * Serum bilirubin >1.5 x ULN (unless due to Gilbert's syndrome)
* Have evidence of any other significant clinical disorder or laboratory finding that, as judged by the investigator, makes it undesirable for the patient to participate in the trial
* Have any evidence of a severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic, or renal disease, active infection (including hepatitis B, hepatitis C, HIV), active bleeding diatheses, or renal transplant)
* Have refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would adversely affect the absorption/bioavailability of the orally administered trial medication
* Any other active malignancy which, in the opinion of the investigator would limit the ability of the patient to complete the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Phase I: The occurrence/non-occurrence of dose limiting toxicities (DLTs) in the trial defined assessment period | During cycle 1 (each cycle is 28 days)
Phase II: Response to treatment as measured by morphological response | At the end of cycle 1 (each cycle is 28 days)
Phase II: For patients with CNS involvement only response to treatment as measured by clearance of Cerebral Spinal Fluid (CSF) blasts | At the end of cycle 1 (each cycle is 28 days)

SECONDARY OUTCOMES:
Phase I & II: The occurrence of adverse events (AEs) as measured by Common Terminology Criteria for Adverse Events (CTCAE) version 4 | From cycle 1 day 1 until 28 days after End of Treatment (6 cycles, each cycle is 28 days)
Phase I & II: The occurrence of adverse events (AEs) as measured by causality assessment | From cycle 1 day 1 until 28 days after the last treatment (6 cycles, each cycle is 28 days)
Phase I & II: Pharmacokinetic variables of selumetinib in combination with dexamethasone from the concentration time profile measured by area under the plasma concentration versus time curve (AUC) | At cycle 1 day 1, cycle 1 day 4 and cycle 2 day 1 (each cycle is 28 days)
Phase I & II: Pharmacokinetic variables of selumetinib in combination with dexamethasone from the concentration time profile measured by the peak plasma concentration (Cmax) | At cycle 1 day 1, cycle 1 day 4 and cycle 2 day 1 (each cycle is 28 days)
Phase I & II: Pharmacokinetic variables of selumetinib in combination with dexamethasone from the concentration time profile measured by the time to reach peak plasma concentration (Tmax) | At cycle 1 day 1, cycle 1 day 4 and cycle 2 day 1 (each cycle is 28 days)
Phase I & II: Pharmacokinetic variables of selumetinib in combination with dexamethasone from the concentration time profile measured by the time required for the concentration of the drug to reach half of its original value (t1/2) | At cycle 1 day 1, cycle 1 day 4 and cycle 2 day 1 (each cycle is 28 days)
Phase I: Response to treatment assessed by complete remission rate as measured by morphological response in bone marrow (BM) | At the end of cycle 1 (each cycle is 28 days)
Phase I: Response to treatment assessed by complete remission rate as measured by minimal residual disease (MRD) response in BM | At the end of cycle 1 (each cycle is 28 days)
Phase I: For patients with CNS involvement only response to treatment assessed by complete remission rate as measured by clearance of CSF blasts | At the end of cycle 1 (each cycle is 28 days)
Phase I & II: Difference in pharmacokinetics of selumetinib (ΔAUC) when selumetinib is administered as single agent | At cycle 1 day 1, cycle 1 day 4 and cycle 2 day 1 (each cycle is 28 days)
Phase I & II: Difference in pharmacokinetics of selumetinib (ΔAUC) when selumetinib is administered in combination with dexamethasone | At cycle 1 day 1, cycle 1 day 4 and cycle 2 day 1 (each cycle is 28 days)
Phase II: The occurrence/non-occurrence of DLTs in the trial defined assessment period | During cycle 1 (each cycle is 28 days)
Phase II: MRD response in BM | At the end of cycle 1 (each cycle is 28 days)

OTHER OUTCOMES:
Exploratory pharmacodynamic biomarker studies including levels of phosphorylated Extracellular signal-regulated kinase (ERK) by flow cytometry as well as retrospective messenger ribonucleic acid (mRNA) profiling, including Bcl-2-like protein 11 (BIM) | Cycle 1 day 1, cycle 1 day 4 and End of Treatment (6 cycles, each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Menne, Principal Investigator — The Newcastle Hospitals NHS Foundation Trust
Locations (17):
- Rigshospitalet, Copenhagen, Denmark
- Prinses Maxima Centrum Voor Kinderoncologie, Utrecht, Netherlands
- United Kingdom (15):
  - Queen Elizabeth Hospital, Birmingham
  - Birmingham Children's Hospital, Birmingham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Alder Hey Children's Hospital, Liverpool
  - University College Hospital Adult Unit, London
  - University College Hospital Paediatric/Teenage & Young Adult Unit, London
  - King's College Hospital, London
  - Hammersmith Hospital, London
  - Great Ormond Street Hospital, London
  - The Christie Hospital, Manchester
  - Great North Children's Hospital, Royal Victoria Infirmary, Newcastle
  - Freeman Hospital, Newcastle
  - Royal Hallamshire Hospital, Sheffield
  - Department of Paediatric Oncology, Royal Marsden Hospital, Sutton, Sutton
  - Haemato-Oncology Adult Unit, Royal Marsden Hospital, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request. The CRCTU is committed to responsible and controlled sharing of anonymised clinical trial data with the wider research community to maximise potential patient benefit while protecting the privacy and confidentiality of trial participants. Data anonymised in compliance with the Information Commissioners Office requirements, using a procedure based on guidelines from the MRC Methodology Hubs, will be available for sharing with researchers outside of the trials team within 6 months of the primary publication. More detailed information on the CRCTU's Data Sharing Policy and the mechanism for obtaining data can be found on the CRCTU website: https://www.birmingham.ac.uk/research/activity/mds/trials/crctu/index.aspx.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available within 6 months of the primary publication.
Access Criteria: See Plan Description above.

REFERENCES:
- [Background] Menne T, Slade D, Savage J, Johnson S, Irving J, Kearns P, Plummer R, Shenton G, Veal GJ, Vormoor B, Vormoor J, Billingham L. Selumetinib in combination with dexamethasone for the treatment of relapsed/refractory RAS-pathway mutated paediatric and adult acute lymphoblastic leukaemia (SeluDex): study protocol for an international, parallel-group, dose-finding with expansion phase I/II trial. BMJ Open. 2022 Mar 4;12(3):e059872. doi: 10.1136/bmjopen-2021-059872. PMID 35246426
- See also: Trial Website — https://www.birmingham.ac.uk/seludex